CLINICAL TRIAL: NCT04963855
Title: A Two-part, Double-blind, Placebo-controlled, Phase I Study of the Safety and Pharmacokinetics of Single Doses of GT300 in Healthy Subjects
Brief Title: A Phase I Study of GT300 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Generian Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-0101
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Lewy Body Disease
MeSH Terms: conditions — Lewy Body Disease | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT300 (Active Comparator): GT300 capsule given once daily
  Interventions: Drug: GT300
- Placebo (Placebo Comparator): Microcrystalline cellulose capsule given once daily
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: GT300 — SIngle oral dose
  Arms: CT300
Drug: Microcrystalline cellulose — placebo
  Arms: Placebo

SUMMARY:
Descriptive safety and pharmacokinetics of GT300, exploratory biomarker effects for the evaluation of the effect of GT300 on the autophagy-lysosomal pathway (ALP), food effect on PK and fasting effect on biomarkers.

DETAILED DESCRIPTION:
This is a two-part study to be conducted under double-blind conditions. Part A will be conducted first and completed before Parts B is conducted.

Part A is a single ascending dose evaluation of GT300 under double blind conditions in a population of healthy male and female subjects. Part B will be conducted once follow-up of the last cohort Part A has been conducted. On each study day in which drug is administered, dosing will be "staggered". Additionally, during Part A, a "sentinel" group comprising 1 active and 1 placebo subject will be dosed approximately 24 hours prior to dosing the remaining 6 subjects in group 1 (5 active, 1 placebo).

Conduct of the study including clinical evaluation of subjects (up to the safety review meeting) will be under double-blind conditions. Progress from one cohort to the next will be contingent on satisfactory review of the safety and other data from each cohort.

Part B is a single dose evaluation of the effect of food and prolonged fasting on the GT300 PK and biomarkers. The dose of GT300 will be equal to, or less than the maximum dose evaluated in Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (non-lactating) subjects age 18 to 55 inclusive.
2. Good general health, with no significant medical history. Subjects must have no clinically significant abnormalities on physical examination at screening, and/or before administration of the initial dose of study drug.
3. Body weight ≥ 50 kg at the screening visit.
4. Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive.
5. Has laboratory values (clinical chemistry, hematology and coagulation) within the normal reference range. Deviations from this range may be acceptable if they are considered 'not clinically significant' (NCS) by the PI.
6. Women of childbearing potential may be enrolled if one of the following criteria applies:

   1. Must be using an effective form of contraception (e.g., oral contraceptives, vaginal ring, IUD, injected or implanted hormonal contraception) for at least one month prior to study entry, must have maintained a normal menstrual pattern for the three months prior to study entry and have a negative pregnancy test (urine) at the time of admission to the unit. Women must be willing to continue this contraception for 90 days following administration of study drug. Their male partner should use a condom.
   2. Is sexually abstinent (Investigator judgement)
   3. Is monogamous with a vasectomized (by history; see section 4.2) months prior)
   4. Is postmenopausal (i.e., amenorrheic for at least 12 months prior to dosing and demonstrating FSH (follicle-stimulating hormone) consistent with post-menopausal state
   5. negative pregnancy test (urine) both at Screening (serum) and Day -1(urine)
   6. Is surgically sterilized (confirmed by medical record review)
   7. Has had a total hysterectomy a minimum of 3 months prior to dosing on Day 1 (confirmed by medical record review)
7. Males who are sexually abstinent may be enrolled or, if sexually active, may be enrolled if one of the following criteria applies:

   1. Has had a vasectomy (>3 months prior to dosing, by history; see section 4.2)
   2. Using condoms and whose partner is using an acceptable form of contraception (IUD, oral contraceptives, birth control patch or vaginal ring, injectable or implanted contraceptives, or tubal ligation [surgical sterilization]) from Day -1 to 90 days after study drug administration; using condom with same sex partner
8. Is a light smoker (on average <10 cigarettes/week) or non-smoker and must not have used any nicotine products within one months prior to dosing. Able and willing to attend the necessary visits to the study center.

Exclusion Criteria:

1. Blood donation or recipient of blood transfusion in previous 12 weeks.
2. History of clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases. Cardiovascular history should include assessment of risk factors for Torsades de Pointes Risk (e.g., heart failure, pulmonary edema, cardiomyopathy, hypokalemia, hypomagnesemia, or hypocalcemia, or family history of Long QT Syndrome, syncope or sudden death).
3. History of neoplastic disease (with the exception of adequately treated non-melanomatous skin carcinoma).
4. Mentally or legally incapacitated (e.g., has significant emotional problems at the time of Screening Visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder within the last 5 years).
5. Fever (body temperature >38C) or symptomatic viral/bacterial infection or use of antibi-otics within 2 weeks prior to Screening.
6. Resting blood pressure (semi-recumbent) (BP) >140/90 mmHg or heart rate (HR) outside the range 40 to 100 beats per minute at Screening and at Day -1.
7. Clinically significant abnormality on ECG performed at the Screening Visit or prior to administration of the initial dose of study drug. (Sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or bundle branch block.
8. Clinically significant laboratory abnormalities including: Impaired renal function (estimated creatinine clearance (CrCl) of <80 mL/minute based on Creatinine Clearance Value as determined by the clinical chemistry laboratory. Additionally, subjects with elevated unconjugated bilirubin consistent with Gilbert's Syndrome are excluded.
9. Positive test for hepatitis C antibody, hepatitis B surface antigen, or human immunodefi-ciency virus (HIV) antibody at Screening.
10. Participants with a positive toxicology screening panel (urine test including qualitative identi¬fication of barbiturates, tetrahydrocannabinol, amphetamines, benzodiazepines, opiates, cocaine and cotinine).
11. Participants with a history of substance abuse or dependency or history of recreational IV drug use (by self-declaration).
12. Alcohol consumption >21 alcohol units per week. (One unit of alcohol is 10 ml, information on calculation the content of drinks is provided at: the "alcohol.gov.au" website.
13. Unable to refrain from or anticipates the use of any medications, including prescription and non-prescription drugs and herbal remedies (such as St. John's Wort [Hypericum perforatum]), beginning 14 days (or 5 half-lives, whichever is longer) before administration of the initial dose of study drug and continuing throughout the study until the follow-up visit. There may be certain medications that are permitted at the discretion of the Investigator and Sponsor (including paracetamol/acetaminophen, multi-vitamin preparations, medications for the treatment of AEs following administration of study drug and immunizations, in particular any one of the COVID-19 vaccines currently in use in AU).
14. Subjects who are unlikely to comply with the study protocol or, in the opinion of the inves-tigator, would not be a suitable candidate for participation in the study.
15. Have participated in any other investigational drug trial within 30 days of dosing in the present study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-08-23 (Estimated); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic | 8 days
  Cmax

IPD SHARING:
Plan to Share IPD: No